CLINICAL TRIAL: NCT04958265
Title: A Phase III, Multicenter, Single-Arm Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Crovalimab in Pediatric Patients With Atypical Hemolytic Uremic Syndrome (aHUS)
Brief Title: A Study Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Crovalimab in Pediatric Participants With Atypical Hemolytic Uremic Syndrome (aHUS)
Acronym: COMMUTE-p
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO42354; 2020-002437-15 (EudraCT Number); 2023-505638-82-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Atypical Hemolytic Uremic Syndrome
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crovalimab (Experimental): Participants will be enrolled in three cohorts: [1] Naive Cohort - participants who have not been previously treated with complement inhibitor therapy; [2] Switch Cohort - participants who switch to crovalimab from another C5 inhibitor and [3] Pretreated Cohort (includes C5 SNP (Single Nucleotide Polymorphism) participants) - participants who received treatment with another C5 inhibitor and subsequently discontinued it.
  Interventions: Drug: Crovalimab

INTERVENTIONS:
Drug: Crovalimab — Crovalimab will be administered at a dose of 1000 mg intravenously (IV) (for participants weighing => 40 to <100 kg) or 1500 mg IV (for participants weighing >=100 kg) on Week 1 Day 1. On Week 1 Day 2 and on Weeks 2, 3 and 4, crovalimab will be administered at a dose of 340 mg subcutaneously (SC). On Week 5 and Q4W thereafter, it will be administered at a dose of 680 mg SC (for participants weighing => 40 to <100 kg) or 1020 mg SC (for participants weighing >=100 kg). Enrollment of participants weighing <40 kg will be staggered using two weight-based dose confirmation groups (Group 1 participants weighing >=20 kg to <40 kg, followed by Group 2 participants weighing >=5 kg to <20 kg). All participants will receive an initial IV loading dose, which will be followed by SC dosing at either Q2W or Q4W intervals (depending on body weight), until study completion.

SUMMARY:
This study aims to evaluate the efficacy and safety of crovalimab in pediatric participants with aHUS.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >= 5 kg at screening.
* Vaccination against Neisseria meningitis serotypes A, C, W, and Y; vaccination against serotype B, according to national vaccination recommendations.
* Vaccination against Haemophilus influenzae type B and Streptococcus pneumoniae, according to national vaccination recommendations.
* For patients continuing to receive other therapies concomitantly with crovalimab (e.g., immunosuppressants, corticosteroids, mammalian target of rapamycin inhibitor (mTORi), or calcineurin inhibitors): stable dose for >=28 days prior to screening and up to the first crovalimab administration.
* For female participants of childbearing potential: an agreement to remain abstinent or use contraception.
* Participants with a prior kidney transplant are eligible if they have a known history of complement-mediated aHUS prior to the kidney transplant.
* Onset of initial TMA presentation within 28 days prior to the first dose of crovalimab (for Naive Cohort only).
* Documented treatment with either eculizumab or ravulizumab (for Switch Cohort only).
* Clinical evidence of response to a C5 inhibitor (for Switch Cohort only).
* Poorly controlled TMA following treatment with another C5 inhibitor (for C5 SNP participants in the Pretreated Cohort only).
* Known C5 polymorphism (for C5 SNP participants in the Pretreated Cohort only).

Exclusion Criteria:

* TMA associated with non-aHUS related renal disease.
* Positive direct Coombs test.
* Chronic dialysis within 90 days prior to first crovalimab administration , and /or end stage renal disease
* Identified drug exposure-related TMA.
* Presence or history of a condition that could trigger TMA, such as malignancy, bone marrow or organ transplant (other than kidney transplant) or autoimmune disease.
* History of a kidney disease, other than aHUS.
* History of Neisseria meningitidis infection within 6 months of study enrollment.
* Known or suspected immune deficiency (e.g., history of frequent recurrent infections).
* Positive HIV test.
* Active systemic bacterial, viral, or fungal infection within 14 days before first crovalimab administration.
* Presence of fever (>= 38°C) before the first crovalimab administration (If fevers are solely due to the underlying aHUS pathology, and there is no evidence or suspicion of a systemic infection, participants may enroll).
* Multi-system organ dysfunction or failure.
* Recent intravenous immunoglobulin (IVIg) treatment.
* Pregnant or breastfeeding or intending to become pregnant.
* Participation in another interventional treatment study with an investigational agent or use of any experimental therapy within 28 days of screening or within five half lives of that investigational product, whichever is greater.
* Recent use of tranexamic acid.
* Current or previous treatment with a complement inhibitor (for Naive Cohort only).
* First initiation of plasma exchange/plasma infusions (PE/PI) should not be more than 28 days prior to first crovalimab administration (for Naive Cohort only).
* Last PE/PI completed less than 2 hours prior to first crovalimab administration (for Naive Cohort only).
* Receiving PE/PI within 8 weeks of the first crovalimab administration (Switch Cohort only).
* Normalization of serum creatinine values at baseline (<97.5th percentile for age), (for Naive Cohort only).
* Positive for active Hepatitis B and/or C infections (HBV/HCV) (for Switch Cohort and switching C5 SNP Pretreated Cohort participants who recently received C5 inhibitor treatment).
* Cryoglobulinemia at screening (for Switch Cohort and C5 SNP Cohort participants who recently received C5 inhibitor treatment).
* Diagnosis of a condition leading to non-aHUS TMA: Thrombotic Thrombocytopenic Purpura (TTP), Shiga Toxin producing Escherichia Coli (STEC)-TMA, Pneumococcal HUS, TMA secondary to cobalamin C defect (as demonstrated by either increased total blood homocysteine levels or MMACHC gene mutation) and TMA related to Diacylglycerol kinase ε (DGKE) nephropathy.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2029-05-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with complete TMA response (cTMAr) (Naive Cohort only) | Baseline up to Week 25 (after 24 weeks on treatment)

SECONDARY OUTCOMES:
Change from Baseline in Dialysis Status | Baseline up to Week 25 (after 24 weeks on treatment)
Change in Estimated Glomerular Filtration Rate (eGFR) (Naive and Switch Cohorts) | Baseline up to Week 25 (after 24 weeks on treatment)
Percentage of Participants with Change from Baseline in Chronic Kidney Disease (CKD) stage (Naive and Switch Cohorts) | Baseline up to Week 25 (after 24 weeks on treatment)
Observed Value in Platelet Count (Naive and Switch Cohorts) | Baseline up to Week 25 (after 24 weeks on treatment)
Observed Value in Lactate Dehydrogenase (LDH) (mg/dL) (Naive and Switch Cohorts) | Baseline up to Week 25 (after 24 weeks on treatment)
Observed Value in Hemoglobin (mg/dL) (Naive and Switch Cohorts) | Baseline up to Week 25 (after 24 weeks on treatment)
Change from Baseline in Platelet Count (Naive and Switch Cohorts) | Baseline up to Week 25 (after 24 weeks on treatment)
Change from Baseline in Lactate Dehydrogenase (LDH) (mg/dL) (Naive and Switch Cohorts) | Baseline up to Week 25 (after 24 weeks on treatment)
Change from Baseline in Hemoglobin (mg/dL) (Naive and Switch Cohorts) | Baseline up to Week 25 (after 24 weeks on treatment)
Percentage of Participants with Platelet Count >= LLN (Naive Cohort only) | Baseline up to Week 25 (after 24 weeks on treatment)
Percentage of Participants with Normalisation of LDH (i.e., =< Upper Limit Normal (ULN)) (Naive Cohort only) | Baseline up to Week 25 (after 24 weeks on treatment)
Percentage of Participants with >=25% decrease in Serum Creatinine (Naive Cohort only) | Baseline up to Week 25 (after 24 weeks on treatment)
Time to complete TMA response (cTMAr) (Naive Cohort only) | Up to 8 years
Duration of complete TMA response (cTMAr) (Naive Cohort only) | Up to 8 years
Percentage of Participants with ongoing complete TMA response (cTMAr) (Naive Cohort only) | At Week 25
Percentage of Participants with maintained TMA control (mTMAc) (Switch Cohort only) | Baseline through Week 25 (after 24 weeks on treatment)
Percentage of Participants with Adverse Events (AEs) | Up to 8 years
Percentage of Participants with Injection-Site Reactions, Infusion-Related Reactions, Hypersensitivity, Malignant Hypertension (including malignant renal hypertension) and Infections (including meningococcal meningitis) | Up to 8 years
Percentage of Participants with Adverse Events (AEs) leading to Study Drug Discontinuation | Up to 8 years
Percentage of Participants with Clinical Manifestations of Drug-Target-Drug Complex (DTDC) formation amongst participants who switched to crovalimab treatment from eculizumab/ravulizumab treatment (Switch Cohort and switching Pretreated participants) | Up to Week 25
Serum Concentrations of Crovalimab over time | Up to 8 years
Prevalence of Anti-Crovalimab Antibodies at Baseline | Baseline
Percentage of Participants with Anti-Crovalimab Antibodies | Up to 8 years
Observed value of Pharmacodynamic Markers (CH50, Free/Total C5) | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Nebraska, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UT Health Science Center, San Antonio, Texas
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Inst. Da Criança- Faculdade de Medicina Usp, São Paulo, São Paulo, Brazil
- CHU Sainte-Justine, Montreal, Quebec, Canada
- China (3):
  - Peking University First Hospital, Beijing
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - The children's hospital , Zhejiang university school of medicine, Hangzhou
- France (2):
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Gh Necker Enfants Malades, Paris
- India (3):
  - Institute of Kidney Diseases and Research Centre, Ahmedabad, Gujarat
  - Medanta-The Medicity, Gurgaon, Haryana
  - All India Institute Of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
- Japan (2):
  - Aichi Children?s Health and Medical Center, Aichi
  - Chiba Children's Hospital, Chibashi, Chibaken
- Hospital de Especialidades Puerta de Hierro S.A de C.V., Zapopan, Mexico
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing